CLINICAL TRIAL: NCT03859349
Title: Routine Systematic Sampling vs. Targeted Sampling of Mediastinal Lymph Nodes Prior to Lung Cancer Treatment: A Feasibility Randomized Controlled Trial
Brief Title: The Canada Lymph Node Score: A Feasibility Randomized Controlled Trial
Acronym: CLNS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: St. Joseph's Healthcare Hamilton (Other)
Collaborators: McMaster University (Other)
Responsible Party: Principal Investigator, Wael Hanna, Head of Endoscopy Services, Thoracic Surgeon, St. Joseph's Healthcare Hamilton
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: sjhhclns_5829
Record Dates: First submitted 2019-02-19; First posted 2019-03-01 (Actual); Last update posted 2020-06-16 (Actual); Status verified 2020-06

CONDITIONS: Non Small Cell Lung Cancer
Keywords: Endobronchial Ultrasound; Diagnostic Imaging; Feasibility; Randomized Controlled Trial; Clinical N0-N1 Disease
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Intervention Model Description: All participants who provide consent for participation and who fulfil eligibility criteria will be randomized with a unique randomization sequence derived from the random permuted block design (with blocks of varying sizes) in a 1:1 ratio. Participants will randomized to either Systematic Sampling (Control) or Targeted Sampling (Experimental).
Who Masked: Participant
Masking Description: Trial participants will remain blinded to their randomized treatment. Additionally, the biostatistician performing the analysis will be blinded as to which intervention arm participants were allocated to, as the group allocations will be coded as Group A and Group B. Provided this is an endoscopic trial, endoscopist blinding will not be feasible. Nonetheless, all patients deemed surgical candidates after EBUS will have their pathology compared to EBUS staging in order to ensure appropriate diagnosis. Pathologists performing such pathology report will be blinded to which intervention arm participants are allocated to.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Systematic Sampling (Active Comparator): Patients will undergo systematic sampling of lymph node stations in the mediastinum with a minimum sampling of 3 stations: 4R, 4L and 7, as is the standard of care. Other stations may be included at the endoscopist's discretion. CLNS is not used for this arm.
  Interventions: Diagnostic Test: Systematic Sampling
- Selective Targeted Sampling (Experimental): Patients will first undergo endosonographic assessment of 3 mediastinal lymph node stations (i.e. 4R, 4L, and 7) using the four criteria of the CLNS. Lymph node stations that exhibit a CLNS >1/4 will be biopsied as is standard of care. Lymph node stations with CLNS ≤ 1/4 will be marked as "not requiring biopsy" but will be biopsied nevertheless, so that there is no deviation from the standard of care. Other stations may be included at the endoscopist's discretion.
  Interventions: Diagnostic Test: Selective Targeted Sampling

INTERVENTIONS:
Diagnostic Test: Selective Targeted Sampling — After CLNS assessment, patients with proven malignant mediastinal lymph nodes will be referred for chemoradiation and patients with proven benign mediastinal lymph nodes will undergo surgical resection as per standard of care guidelines. Final pathology from the resected specimen will be considered the gold standard for analysis of sensitivity and specificity.
  Other Names: STS; CLNS
  Arms: Selective Targeted Sampling
Diagnostic Test: Systematic Sampling — Following routine biopsy of lymph nodes, patients with proven malignant mediastinal lymph nodes will be referred for chemoradiation and patients with proven benign mediastinal lymph nodes will undergo surgical resection as per standard of care guidelines. Final pathology from the resected specimen will be considered the gold standard for analysis of sensitivity and specificity.
  Other Names: Routine Mediastinal Staging; SS
  Arms: Systematic Sampling

SUMMARY:
For patients diagnosed with early stage Non-Small Cell Lung Cancer (NSCLC) on preoperative computerized tomography (CT) and positron emission tomography (PET) scans, surgical resection is usually the preferred method of treatment. However, to be eligible for surgery, current guidelines require that the cancer has not spread to the lymph nodes in the chest cavity. To evaluate these lymph nodes, the standard of care is to undergo an endobronchial ultrasound (EBUS) procedure, where all the visible lymph nodes in the chest are biopsied (sampled) with a needle. Unfortunately, these biopsies are often inconclusive, especially in patients who have no evidence of mediastinal lymph node spread on pre-operative imaging. Currently, the standard of care mandates that inconclusive biopsies should be repeated, either through another EBUS, or through more invasive procedures. Repeat inconclusive biopsies are oftentimes inconclusive as well; leading to a vicious cycle of inconclusive results, a delay in treatment, morbidity for the patient, and increased costs to the healthcare system. To circumvent this issue, the investigators have developed, validated and published a 4-point score, the Canada Lymph Node Score (CLNS), which uses four features observed during EBUS to predict whether the cancer has spread to the lymph nodes or not. Research has demonstrated that lymph nodes which appear benign on both CT and PET scan that also have a CLNS of ≤1/4 are almost certainly benign. As such, it is believed that these "triple normal" lymph do not require biopsy (or repeat biopsy).

The investigators are challenging the current standard of care in lung cancer, which mandates that all the lymph nodes in the chest need to be biopsied (i.e. Systematic Sampling) before surgery, by proposing that triple normal lymph nodes can be omitted, and only those with cancer potential should be biopsied (i.e. Targeted Sampling).To prove this hypothesis, a randomized controlled trial comparing Systematic Sampling to Targeted Sampling is required. A feasibility trial is proposed to determine whether this large-scale randomized trial will be possible.

ELIGIBILITY:
Inclusion Criteria:

* Referred to have EBUS for staging of confirmed or suspected NSCLC
* Completed both a CT and PET scans
* cN0-cN1 disease indicated on CT and PET scans

Exclusion Criteria:

* Patients with cN0 disease, peripheral tumours and tumours < 2 cm in diameter (they do not require staging)
* Evidence of cN2 disease or higher on CT and PET scan

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2019-05-06 (Actual); Primary Completion 2020-03-02 (Actual); Study Completion 2020-06-08 (Actual)

PRIMARY OUTCOMES:
Recruitment Rate | 1 Year
  Minimum acceptable recruitment rate is 70%
Procedure Length | 1 Day
  Calculated in minutes. Recorded for both treatment arms.
Diagnostic Accuracy | 1 Year
  The proportion of patients in whom the treatment (CLNS or biopsy) yielded the same diagnosis as the pathology report out of the total number of patients that have received the treatment. Recorded for both treatment arms.

SECONDARY OUTCOMES:
Prevalence of Each Possible CLNS | 1 Year
  The CLNS has five possible scores: 0/4, 1/4, 2/4, 3/4 and 4/4. The number of lymph nodes with each score will be recorded for the Experimental Arm (Targeted Sampling).
Frequency of Biopsies | 1 Year
  Number of times lymph nodes had to be sampled with a transbronchial needle per EBUS procedure. Recorded for both treatment arms.
Percent of Inconclusive Biopsies | 1 Year
  Number of biopsies that provided an inconclusive diagnosis out of total number of biopsies obtained. Recorded for each treatment arm.
Adverse Events | 1 Year
  Number of AEs has classified by the Ottawa TM&M System
Accrual Period | 1 Year
  Duration of time to reach sample size

CONTACTS AND LOCATIONS:
Overall Officials: Waël C Hanna, MDCM, MBA, FRCSC, Principal Investigator — St. Joseph's Healthcare Hamilton / McMaster University
Locations (1):
- St. Joseph's Healthcare Hamilton, Hamilton, Ontario, Canada

REFERENCES:
- [Derived] Sullivan KA, Farrokhyar F, Leontiadis GI, Patel YS, Churchill IF, Hylton DA, Xie F, Seely AJE, Spicer J, Kidane B, Turner SR, Yasufuku K, Hanna WC. Routine systematic sampling versus targeted sampling during endobronchial ultrasound: A randomized feasibility trial. J Thorac Cardiovasc Surg. 2022 Jul;164(1):254-261.e1. doi: 10.1016/j.jtcvs.2021.11.062. Epub 2021 Dec 4. PMID 35031139